CLINICAL TRIAL: NCT02892175
Title: Can the Vascular Physician Sensitize Patients to Redaction of Advance Directives on End of Life?
Acronym: DIRFIN
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DIRFIN
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: End of Life
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Advance Directives on End of Life — after information transmitted orally by the doctor (Dr P.Priollet) and agreement of the patient to participate, patients will be interviewed (Questionary) and data collected during visits to consultations City office of Dr. Priollet by Dr. Priollet assisted by Mrs. Helena Sanson (internal medicine), anonymized and handled within the vascular medicine department of Dr. Priollet to GHPSJ.

SUMMARY:
The Leonetti law of 22 April 2005 on the rights of patients at end of life provides the opportunity for "all adults" to write advance directives in case she would one day be "unable to express their will." If this right is enshrined in the hospitalized patient's charter, brought to the attention of any patient entering a hospital, the fact remains that only 2.5% of the deceased have written advance directives (study National Institute of demographic studies published in 2012).

Moreover, according Régis Aubry, a researcher at the observatory on the end of life, the conditions of the end of life are insufficiently discussed with patients and their families and can lead to difficult situations conflicting view. Now, thinking about advance directives should allow an exchange on the conditions of the end of life desired by patients.

Sicard report of December 2012 concluded that such legislation is known neither patients nor doctors. This is the first obstacle to its use, even if major psychological barriers exist both in patients that their doctors.

It is in this context that Valls government asked MM. Claeys and Leonetti to propose a new bill on the subject. The bill provides that advance directives will no longer be valid for 3 years, but until changed or until the patient's death, and they can be invoked against doctors except emergency or illegality. In addition, to complete the bill, the Ministry of Health commissioned the National Health Authority (HAS) writing a form of advance directives, as well as a doctor's information guide and patient on the subject. The working group is chaired by Professor Sicard. Among the recommendations made to physicians (and by extension health professionals), the investigators accept that talk of advance directives as often as possible and as early as possible, even in the absence of commitment in the short or medium term prognosis .

DETAILED DESCRIPTION:
Main objective / secondary:

Feasibility of addressing the topic of advance directives (% of patients agreeing to answer the questionnaire) during vascular medicine clinic in town.

Assessing preferences for editorial context to enable to present the project in optimal circumstances.

Assess felt an evolution of the doctor-patient relationship by patients in the context of advance directives.

Assess the reactions according to the characteristics of the study population to help develop different "profiles" and adapt the introduction of the topic of advance directives.

Methodology :

Design: prospective, single-center, non-interventional kind opinion survey Study duration: 6 months

Acquisition of data:

The characteristics of the population obtained will be studied to try to understand the feelings of patients, to better target patients to talk to about advance directives in vascular medicine and evaluate some extent if the topic of advance directives contributes to "modernize "the doctor-patient relationship.

* List of data gathered: cf. attached questionnaire
* Statistical analysis: local management (GHPSJ) from the patient profile
* Anonymity of data: an identifier for each subject will be awarded (first name and surname - year of birth) and the data will be entered on a computer file which will be sent to the statistician in charge of analyzing the GHPSJ site. There will be no personally identifiable data exchange.

Development of the study:

* Describe how the study: after information transmitted orally by the doctor (Dr P.Priollet) and patient's consent to participate, patients will be interviewed (attached schedule) and data gathered during consultations of office visits to Dr. Priollet city by Dr. Priollet assisted by Hélène Samson (internal medicine), anonymized and handled within the vascular medicine department of Dr. Priollet to GHPSJ.
* Expected duration of patient recruitment: 3 months
* Number of patients to recruit 100 patients, 15 minutes per patient. At all times patients can freely return to the subject in subsequent consultations with Dr. Priollet.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients already followed in the vascular medicine department

Exclusion Criteria:

* Patients refusing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive patients already followed in the vascular medicine department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the number of patients agreeing to answer the questionary | Day 1

SECONDARY OUTCOMES:
Assessment of the felt of the patient on a scale | Hour +1
  Assess of felt an evolution of the doctor-patient relationship by patients in the context of advance directives. A scale is used from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided